CLINICAL TRIAL: NCT02506621
Title: Randomised ELR Monitoring Against Permanent Pacemaker in Atrial Fibrillation
Brief Title: ELR Monitoring Against Permanent Pacemaker in Atrial Fibrillation
Acronym: REMAP-AF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eastbourne General Hospital (Other)
Responsible Party: Principal Investigator, Neil Sulke, Dr, Eastbourne General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: REMAP-AF version 1.0
Record Dates: First submitted 2015-07-16; First posted 2015-07-23 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ELR monitoring (Experimental): Single arm study. All participants with existing permanent dual chamber pacemakers will be monitored with 5 different Loop recorder devices for a 2 week period to assess there sensitivity and specificity in detecting AF burden. The devices used will be
  1. R test
  2. Nuubo
  3. TECHNOMED pocket ECG
  4. ZIO xt patch
  5. MoMe
  Interventions: Device: R test; Device: Nuubo; Device: TECHNOMED pocket ECG; Device: ZIO xt patch; Device: MoMe

INTERVENTIONS:
Device: R test
Device: Nuubo
Device: TECHNOMED pocket ECG
Device: ZIO xt patch
Device: MoMe

SUMMARY:
Randomised crossover study comparing the sensitivity and specificity of 5 External loop recorders in detecting pacemaker detected Atrial fibrillation burden.

DETAILED DESCRIPTION:
The purpose of the study is to compare the diagnostic accuracy of the ZIO xt , MoMe, TECHNOMED pocket ECG and Nuubo to the R-test, our current standard clinical practice, in detection of AF burden, in patients with history of Paroxysmal Atrial Fibrillation and have a dual chamber pacemaker or ICD in situ, with sensitivity and specificity of AF detection calculated from the implanted pacemaker monitored beat to beat holters.

ELIGIBILITY:
Inclusion Criteria:

* History of Atrial Fibrillation
* Dual chamber pacemaker with advanced holter arrhythmia diagnostics

Exclusion Criteria:

* Previous AV node ablation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-09; Primary Completion 2015-12 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity in detection of pacemaker detected AF burden in comparison to R-test | 14 weeks
  Sensitivity and specificity of ZIO xt patch, MoMe, TECHNOMED pocket ECG AND Nuubo in detection of pacemaker detected AF burden in comparison to R-test.
  Sensitivity and sepcificity will be determined by the percentage of pacemaker detected AF episodes that have been detected by each ELR device.

SECONDARY OUTCOMES:
proportion of pacemaker detected tachyarrhythmias detected in comparison to R-test | 14 weeks
  Proportion of pacemaker detected tachyarrhythmias detected by the ZIO xt patch, MoMe, TECHNOMED pocket ECG and Nuubo in comparison to R-test
Total wear time in comparison to R-test | 14 weeks
  Total wear time of the ZIO xt patch, MoMe, TECHNOMED pocket ECG and Nuubo in comparison to R-test
Proportion of symptomatic arrhythmias detected in comparison to R-test | 14 weeks
  Proportion of symptoms secondary to arrhythmias detected by the ZIO xt patch, MoMe, TECHNOMED pocket ECG and Nuubo compared to R-Test
Cost effectiveness in detection of arrhythmias in comparison to R-test | 14 weeks
  Cost-effectiveness of ZIO xt patch, MoMe, TECHNOMED pocket ECG and Nuubo in detection of arrhythmia in comparison to R-Test

OTHER OUTCOMES:
User satisfaction in interpretation of reports compare | 14 weeks
  Ease of interpretation of results summary derived by device software - validated by questionnaire provided to junior & senior Cardiologists and junior & senior Physiologists
Participant feedback on device tolerability assessed by Visual Analogue Score (VAS) questionnaire | 14 weeks
  Participant feedback on device tolerability assessed by Visual Analogue Score (VAS) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Neil Sulke, DM, FRCP, Principal Investigator — Eastbourne General Hospital